CLINICAL TRIAL: NCT00552708
Title: A Randomized, Open-label, Single-dose, Crossover Study to Demonstrate the Bioequivalence of the Final Fixed Dose Combination (FDC) Formulation (COREG CR & Lisinopril) to COREG CR & ZESTRIL Employed in the Phase III Factorial Study
Brief Title: A Study Investigating the Bioequivalence of the Fixed Dose Combination of COREG CR to COREG CR and ZESTRIL.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CFD108412
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Hypertension
Keywords: COREG CR
MeSH Terms: conditions — Hypertension | interventions — Carvedilol; Lisinopril

INTERVENTIONS:
Drug: COREG CR
Drug: Lisinopril
  Other Names: COREG CR

SUMMARY:
This study will be a randomized study investigating the bioequivalence of COREG CR to its components, COREG and Lisinopril (ZESTRIL). PK samples will be obtained throughout the study to investigate the PK of COREG CR FDC to COREG and Lisinopril

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females of non-child bearing potential who are between 18 to 55 years of age, inclusively
* Body weight > 60 kg (132 lbs) and body mass index (BMI) between 19 and 33

Exclusion criteria:

* Any clinically relevant abnormality identified on the screening history, physical or laboratory examination, or any other medical condition or circumstance making the volunteer unsuitable for participation in the study.
* Subjects who metabolize carvedilol poorly based on CYP2D6 genotyping as determined at screening.
* Treatment with any prescription or non-prescription drugs (including vitamins, herbal and dietary supplements, as well as grapefruit-containing products) within 7 days or 5 half-lives prior to first dose of study medication and until the end of the study. Treatment with any prescription drugs that are CYP2D6 inhibitors within 14 days prior to the first dose of study medication until the end of the study. Excluded from this list is acetaminophen at doses of ≤ 2 grams/day.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding Day 1 of Session 1.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of regular alcohol consumption exceeding 7 drinks/week for women or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening.
* Positive urine drug screen (UDS) including alcohol at screening. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* Urine Na/creatinine ratio < 0.1 meq/mg.
* Positive for Hepatitis B surface antigen or HIV.
* Women of child-bearing potential.
* Resting heart rate of ≤ 50 beats per minute (bpm) at screening.
* Any abnormalities as defined in the protocol on 12-lead ECG during screening
* Documented history of low blood pressure (average SBP ≤ 110 mm Hg and/or DBP ≤50 mm Hg) or blood pressure below these values at time of screening.
* Orthostatic hypotension diagnosed at screening (orthostatic hypotension will be defined as a reduction in systolic blood pressure of 20 mmHg or more and/or a reduction in diastolic blood pressure of 10 mmHg or more for standing vs. supine measurements.
* Donation of blood in excess of 500 mL within a 56 day period, including ~478 mL of blood drawn during this study.
* History of asthma, COPD and/or hypersensitivity to β-adrenergic blocking agents.
* History of sensitivity to heparin, heparin- induced thrombocytopenia, or sensitivity to any of the study medications or components thereof.
* History of anaphylaxis or anaphylactoid reactions or severe allergic responses to drugs.
* History of angioedema.
* Unwillingness or inability to follow the procedures outlined in the protocol or inability to provide written informed consent.
* History of sensitivity to carvedilol, lisinopril, alpha-blockers, beta-blockers or ACE inhibitors.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To establish bioequivalence of the final FDC product (80 mg carvedilol CR/10 mg lisinopril) relative to concomitant dosing of COREG CR (80 mg) and ZESTRIL (10 mg, over encapsulated)throughout the study | throughout the study

SECONDARY OUTCOMES:
To further evaluate the pharmacokinetic profile of the final FDC product. To evaluate the safety and tolerability of single doses of the fixed dose combination at the highest dose strengths of each component throughout the study | throughout the study
plasma levels of carvedilol to determine pharmacokinetic parameters.
plasma levels of lisinopril determine pharmacokinetic parameters.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States